CLINICAL TRIAL: NCT04836234
Title: The Effect of the Chewing Gum in Alleviating Orthodontic Pain After Separator and Initial Arch Wire Placement: A Randomized Clinical Trial
Brief Title: Chewing Gum Effect in Reducing Orthodontic Pain After Separator and Initial Arch Wire Placement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Malaya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DGD170001
Record Dates: First submitted 2020-11-05; First posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Orthodontic Pain
Keywords: Chewing gum, Orthodontic pain

STUDY DESIGN:
Intervention Model Description: Method of randomization using online randomization software. All 108 participants will be randomly allocated into 2 groups with a 1:1 allocation. Participants will be grouped into either group 1 (Intervention group, chewing gum) or group 2 (Control group, no chewing gum given) by using block randomization with block size of 4. Each group will have 54 participants. Concealment of the allocation sequence will be done by concealing the sequence in opaque envelopes.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Blinding of participants is not possible during allocation, treatment and data collection. However, blinding can be done during data processing, analysing and data collection for secondary outcome on appliances failure rate.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): Participants will receive Wrigley Extra Strawberry Flavour Sugar Free Chewing Gum. They will be instructed to chew the gum for pain relief after the separator and initial arch wire placement if required. Chew the gums for 10-12 minutes and as much as they want whenever they feel discomfort or pain. They are free to take any medication when necessary and respond to the questionnaires on the amount of chewing gum and analgesics used.
  Interventions: Other: Wrigley Extra Strawberry Flavour Sugar Free Chewing Gum
- Control group (No Intervention): Participants will not receive any prescription after the separators and initial arch wires placement. They will be specifically asked not to chew chewing gum. As in the intervention group, they can take any medication when they feel necessary and respond to the questionnaires on the amount of analgesics used.

INTERVENTIONS:
Other: Wrigley Extra Strawberry Flavour Sugar Free Chewing Gum — Wrigley Extra Strawberry Flavour Sugar Free Chewing Gum 65g 40 pieces
  Arms: intervention group

SUMMARY:
Pain is the most claimed complaint from orthodontic treatment. Fear of pain has contributed to patients' avoidance of seeking orthodontic treatment, affects patients' compliance to treatment and even becomes the main reason for discontinuing orthodontic treatment. For years, orthodontic patients have reported using analgesics during orthodontic treatment to ease the pain. However, analgesics have many side effects such as allergic reactions, bleeding disorders, gastric ulcers, liver toxicity and their potential influence in slowing down tooth movement. This study aimed to investigate the effectiveness of chewing gums in pain reduction in Malaysian multi-ethnic orthodontic patients and to explore the possibility of chewing gum to be recommended as a suitable substitute for analgesics in our future practice.

DETAILED DESCRIPTION:
Orthodontic treatment have been shown to cause varying degrees of discomforts and pain to the patients. Fear of pain has contributed to patients' avoidance of seeking orthodontic treatment, affect patients' compliance to the treatment and even become a main reason of discontinuing orthodontic treatment. Patients have reported using of analgesic particularly NSAIDS and Paracetamol during orthodontic treatment to ease the pain. However, NSAIDS have been associated with various side effects such as allergic reactions, bleeding disorders and gastric ulcers had raised the concern of orthodontists. Studies on animals have shown that NSAIDS slower the rate of tooth movement, hence affecting orthodontic treatment efficacy. Paracetamol have been reported to cause liver toxicity in the case of over dosage.

The action of chewing the gum can produce forces to temporary displace the teeth sufficiently to allow blood flow through compressed area, preventing the build-up of metabolic products, thus reduce the pain severity. In addition, non-sugared chewing gum has anti-caries effect which is very important to prevent caries formation during orthodontic treatment.

This study aimed to investigate the effectiveness of chewing gum in pain reduction in orthodontic patients and to explore the possibility of chewing gum to be recommended as a suitable substitute for analgesics in future practice.

ELIGIBILITY:
Inclusion Criteria:

1. Patients about to undergo orthodontic treatment with maxillary and mandibular fixed appliances
2. Orthodontic treatment include the extraction of the permanent first or second premolars
3. Age 16 years and above

Exclusion Criteria:

1. Significant medical problem or cleft lip and palate.
2. Pregnant lady
3. Occurrence of using analgesics or antibiotics
4. History of asthma or unstable asthma the last year
5. Oral surgery in the previous 4 weeks

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2019-03-06 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Pain assessment after separators and initial arch wire placement. | At 6 hours after separators and initial arch wire placement.
  Level of pain on the Numerical pain rating scale (NRS)
Pain assessment after separators and initial arch wire placement. | At 24 hours after separators and initial arch wire placement.
  Level of pain on the Numerical pain rating scale (NRS)
Pain assessment after separators and initial arch wire placement. | At 48 hours after separators and initial arch wire placement.
  Level of pain on the Numerical pain rating scale (NRS)

SECONDARY OUTCOMES:
Reported use of chewing gum and analgesics. | Immediately after the separator and archwire placements until up to 6 hours
  Amount of chewing gums and medications consumed after the separator and initial arch wire placement
Reported use of chewing gum and analgesics. | from 6 hours to 24 hours after the separator and archwire placements
  Amount of chewing gums and medications consumed after the separator and initial arch wire placement
Reported use of chewing gum and analgesics. | from 24 hours to 48 hours after the separator and archwire placements
  Amount of chewing gums and medications consumed after the separator and initial arch wire placement
Recorded appliances breakages. | Immediately after the separator and archwire placements until 2 days after the separator and archwire placement
  Frequency of appliances breakages

CONTACTS AND LOCATIONS:
Overall Officials: Siti Adibah Othman, Prof, Study Director — Faculty of Dentistry, University of Malaya; Zamros Yuzadi Mohd Yusof, Prof, Study Director — Faculty Of Dentistry, University of Malaya; Poon Pei San, Principal Investigator — Faculty of dentistry, University of Malaya
Locations (1):
- Postgraduate Orthodontic Clinic, Faculty of Dentistry, University Malaya, Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Benson PE, Razi RM, Al-Bloushi RJ. The effect of chewing gum on the impact, pain and breakages associated with fixed orthodontic appliances: a randomized clinical trial. Orthod Craniofac Res. 2012 Aug;15(3):178-87. doi: 10.1111/j.1601-6343.2012.01546.x. Epub 2012 Jun 22. PMID 22812440
- [Background] Ireland AJ, Ellis P, Jordan A, Bradley R, Ewings P, Atack NE, Griffiths H, House K, Moore M, Deacon S, Wenger N, Worth V, Scaysbrook E, Sandy JR. Comparative assessment of chewing gum and ibuprofen in the management of orthodontic pain with fixed appliances: A pragmatic multicenter randomized controlled trial. Am J Orthod Dentofacial Orthop. 2016 Aug;150(2):220-7. doi: 10.1016/j.ajodo.2016.02.018. PMID 27476354
- [Background] Kehoe MJ, Cohen SM, Zarrinnia K, Cowan A. The effect of acetaminophen, ibuprofen, and misoprostol on prostaglandin E2 synthesis and the degree and rate of orthodontic tooth movement. Angle Orthod. 1996;66(5):339-49. doi: 10.1043/0003-3219(1996)0662.3.CO;2. PMID 8893104
- [Background] Xiaoting L, Yin T, Yangxi C. Interventions for pain during fixed orthodontic appliance therapy. A systematic review. Angle Orthod. 2010 Sep;80(5):925-32. doi: 10.2319/010410-10.1. PMID 20578865
- [Background] Salmassian R, Oesterle LJ, Shellhart WC, Newman SM. Comparison of the efficacy of ibuprofen and acetaminophen in controlling pain after orthodontic tooth movement. Am J Orthod Dentofacial Orthop. 2009 Apr;135(4):516-21. doi: 10.1016/j.ajodo.2007.05.020. PMID 19361739